CLINICAL TRIAL: NCT07385053
Title: Post-Marketing Clinical Follow Up of ESTYME® LIFT in the Correction of Nasolabial Folds
Brief Title: Real-Life Evaluation of the HA Dermal Filler ESTYME® LIFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1905
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Nasolabial Folds, Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aesthetic Treatment for the Correction of Nasolabial Folds. (Experimental)
  Interventions: Device: Injection of the Hyaluronic Acid-Based Dermal Filler ESTYME® LIFT (Now Marketed as ESTYME® FORM).

INTERVENTIONS:
Device: Injection of the Hyaluronic Acid-Based Dermal Filler ESTYME® LIFT (Now Marketed as ESTYME® FORM). — The device will be used under real-life conditions. Following the initial injection session, an optional touch-up may be performed one month after the first injection. A retreatment session may be offered to the patient between 9 and 24 months after the initial injection.

SUMMARY:
The objective of this post-market interventional study is to confirm, under real-life conditions, the safety and performance of a hyaluronic acid-based dermal filler intended for the aesthetic correction of nasolabial folds. The primary question addressed by the study is: How long does the effect of the product last? Following the initial injection session, which includes an optional touch-up planned one month after the first injection, participants will attend a follow-up visit scheduled between 9 and 24 months after the initial treatment. During this visit, patients may receive a retreatment if they wish.

The flexibility of the follow-up window between 9 and 24 months was defined to allow patients to return on their own initiative for retreatment, thereby indicating the end of the effect of the initial injection session. A final follow-up visit is also scheduled at 24 months.

At each visit, the investigator will assess both performance and safety through a clinical examination. In addition, at each follow-up visit, participants will evaluate the aesthetic improvement compared with their pre-injection appearance.

ELIGIBILITY:
Inclusion Criteria:

* Subject seeking an aesthetic procedure defined by the correction of nasolabial folds with Estyme® LIFT (now marketed as ESTYME® FORM).
* Subject who agreed to participate and have signed an informed consent.
* Age: over 18 years old.
* Subject being affiliated to a health social security system.

Exclusion Criteria:

* Patients with a known allergy to hyaluronic acid, lidocaine or amide local anesthetics.
* Patients with porphyria.
* Patients with an autoimmune disorder, or using an immunosuppressant medication.
* Pregnant or breastfeeding women.
* Patients with cutaneous disorders, inflammation or infection (herpes, acne, etc.) at the treatment siteor nearby.
* Patients with bleeding disorders or in patients receiving thrombolytic or anticoagulant treatment.
* Patients with an active or history of streptococcal diseases.
* Children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who returned to their baseline (pre-injection) state, as assessed by the investigator using the 6-point nasolabial fold scale (0 = no wrinkle; 6 = very deep wrinkle). | At each follow-up visit, including the 9-24-month visit and the 24-month visit.

SECONDARY OUTCOMES:
Number of adverse device effects (ADEs) and serious adverse device effects (SADEs) assessed by the investigator. | From the initial injection (day 0) to the end of the follow-up period (24 months).
Injection site reactions (ISR) assessed by the investigator. | Day 0 (after the first injection), Month 1 (after the optional touch-up), and between Month 9 and Month 24 (after the optional retreatment)
Investigator-assessed severity of nasolabial folds using the 6-point scale (0 = no wrinkle, 6 = very deep wrinkle) | Assessments were performed before and after each injection (D0: initial injection; M1: optional touch-up; between M9 and M24: optional retreatment), as well as at each follow-up visit, including the 9-24-month and 24-month visits.
Aesthetic change, as assessed by the subject compared with baseline, using the 5-point Global Aesthetic Improvement Scale (GAIS) from 'worse' to 'very much improved. | At each follow-up visit, including the 9-24-month visit and the 24-month visit.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Médical Saint Jean, Arras
  - Cabinet médical, Lyon
  - Palais de Flore, Lyon

IPD SHARING:
Plan to Share IPD: No